CLINICAL TRIAL: NCT02836613
Title: Pharmacokinetics and Pharmacodynamics of LY2951742 (Galcanezumab) in Healthy Subjects Following Subcutaneous Administration of LY2951742 (Galcanezumab) Solution in a Prefilled Syringe or an Autoinjector
Brief Title: A Study of Galcanezumab in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16203; I5Q-MC-CGAQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2017-12

CONDITIONS: Healthy
MeSH Terms: interventions — galcanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Galcanezumab Reference (Active Comparator): Single dose of 240 milligrams (mg) galcanezumab (LY2951742) administered subcutaneously (SC) by manual prefilled syringe (PFS).
  Interventions: Biological: Galcanezumab
- Galcanezumab Test (Experimental): Single dose of 240 mg galcanezumab (LY2951742) administered SC by autoinjector.
  Interventions: Biological: Galcanezumab

INTERVENTIONS:
Biological: Galcanezumab — Administered SC
  Other Names: LY2951742

SUMMARY:
The main purpose of this study is to evaluate how much galcanezumab gets into the body after it is given as an injection just under the skin by two different devices. This study will measure how much galcanezumab reaches the blood stream and will test how it affects calcitonin-gene related peptide (CGRP) in blood. Information about any side effects that may occur will be collected. The study will last about 20 weeks for each participant. Screening is required within 45 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy as determined by medical history and physical examination
* Have a body mass index (BMI) between 19.0 and 35.0 kilogram per meter square (kg/m²)
* Have clinical laboratory test results within normal reference range for the investigative site, or results with acceptable deviations that are judged to be not clinically significant by the investigator

Exclusion Criteria:

* Have previously completed or withdrawn from this study or any other study investigating galcanezumab, and have previously received galcanezumab
* Have allergies to either humanized monoclonal antibodies, diphenhydramine, epinephrine, or methylprednisolone
* Intend to use over-the-counter or prescription medication within 7 days prior to dosing and during the study (especially systemic glucocorticoids, immunomodulatory drugs, drugs with propensity for dermal reactions, drugs with known hepatic toxicity, etc). Stable doses of hormone replacement therapy (HRT) are allowed for inclusion at the discretion of the investigator
* Have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02-27 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Covance Clinical Research Inc, Daytona Beach, Florida
  - Covance Clinical Research Inc, Evansville, Indiana
  - Covance, Dallas, Texas

REFERENCES:
- [Derived] Stauffer VL, Sides R, Lanteri-Minet M, Kielbasa W, Jin Y, Selzler KJ, Tepper SJ. Comparison between prefilled syringe and autoinjector devices on patient-reported experiences and pharmacokinetics in galcanezumab studies. Patient Prefer Adherence. 2018 Sep 17;12:1785-1795. doi: 10.2147/PPA.S170636. eCollection 2018. PMID 30271122

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open label, randomized, parallel group with study drug administration on Day 1 and up to 20 weeks blood sampling.
Groups:
- Galcanezumab Pre Filled Syringe (PFS): Single dose of 240 mg galcanezumab administered subcutaneously (SC) by manual prefilled syringe.
- Galcanezumab Autoinjector: Single dose of 240 mg galcanezumab administered SC by autoinjector.
Period: Overall Study
Arm/Group | Galcanezumab Pre Filled Syringe (PFS) | Galcanezumab Autoinjector
Started | 80 | 80
Completed | 79 | 77
Not Completed | 1 | 3
Not completed — Accidental drowning | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Galcanezumab Pre Filled Syringe (PFS): Single dose of 240 mg galcanezumab (LY2951742) administered subcutaneously (SC) by manual prefilled syringe.
- Galcanezumab Autoinjector: Single dose of 240 mg galcanezumab (LY2951742) administered SC by autoinjector.
- Total: Total of all reporting groups
Arm/Group | Galcanezumab Pre Filled Syringe (PFS) | Galcanezumab Autoinjector | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.9) | 38.3 (11.5) | 38.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 81
  Male | 40 | 39 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 17 | 31
  Not Hispanic or Latino | 66 | 63 | 129
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 33 | 31 | 64
  White | 43 | 46 | 89
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 80 | 160
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 78.39 (14.34) | 81.61 (13.72) | 80.00 (14.08)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Galcanezumab
Description: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Galcanezumab
Time Frame: 8, 24, 48,96,120,168,216,264,336,504,672,1008,1344,1680,2016,2688 and 3360 hours post dose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Galcanezumab Pre Filled Syringe (PFS) | Galcanezumab Autoinjector
Number analyzed (Participants) | 74 | 75
micrograms per milliliter (ug/mL) | 31.5 (40) | 32.3 (33)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf] of Galcanezumab
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-inf] of Galcanezumab
Time Frame: 8, 24, 48,96,120,168,216,264,336,504,672,1008,1344,1680,2016,2688 and 3360 hours post dose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | Galcanezumab Pre Filled Syringe (PFS) | Galcanezumab Autoinjector
Number analyzed (Participants) | 74 | 75
day*ug/mL | 1170 (35) | 1110 (35)

3. Secondary Outcome: Pharmacodynamics (PD): Maximum Observed CGRP Concentration (Cmax)
Description: Pharmacodynamics (PD): Maximum Observed CGRP Concentration (Cmax)
Time Frame: Pre dose, 24,48,96,120,168,264,336,504,672,1008,1244,1680,2016,2688, and 3360 hours post dose
Population: All participants who received at least 1 dose of study drug and had evaluable Cmax CGRP PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Galcanezumab Pre Filled Syringe (PFS) | Galcanezumab Autoinjector
Number analyzed (Participants) | 74 | 75
nanograms per milliliter (ng/mL) | 3.11 (41) | 3.13 (48)

4. Secondary Outcome: Pharmacodynamics (PD): Area Under the Concentration Versus Time Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration of CGRP (AUC[0-tlast, CGRP])
Description: Pharmacodynamics (PD): Area Under the Concentration Versus Time Curve from Time Zero to Time T, Where T is the Last Time Point with a Measurable Concentration of CGRP (AUC[0-tlast, CGRP])
Time Frame: Pre dose, 24,48,96,120,168,264,336,504,672,1008,1244,1680,2016,2688, and 3360 hours post dose
Population: All participants who received at least 1 dose of study drug and had evaluable AUC[0-tlast, CGRP] PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Galcanezumab Pre Filled Syringe (PFS) | Galcanezumab Autoinjector
Number analyzed (Participants) | 66 | 63
day*ng/mL | 242 (50) | 242 (58)

ADVERSE EVENTS:
Time Frame: up to 8 months
Description: All participants who received at least 1 dose of study drug.
Arm/Group | Galcanezumab Pre Filled Syringe (PFS) | Galcanezumab Autoinjector
All-Cause Mortality (participants affected / at risk) | 1/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 1/80 | 1/80
Other Adverse Events (participants affected / at risk) | 27/80 | 38/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galcanezumab Pre Filled Syringe (PFS) (N=80) | Galcanezumab Autoinjector (N=80)
Drowning (General disorders) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galcanezumab Pre Filled Syringe (PFS) (N=80) | Galcanezumab Autoinjector (N=80)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 2 (3) | 3 (3)
Injection site erythema (General disorders) | 2 (2) | 4 (6)
Injection site induration (General disorders) | 1 (1) | 2 (3)
Injection site pain (General disorders) | 2 (2) | 10 (14)
Injection site pruritus (General disorders) | 1 (1) | 2 (3)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 6 (6)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 1 (2)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 9 (11)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT02836613/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT02836613/SAP_001.pdf